CLINICAL TRIAL: NCT01347892
Title: Post Market, Longitudinal Data Collection Study of Articular Cartilage Lesions in the Ankle Treated With DeNovo(R) NT Natural Tissue Graft
Brief Title: DeNovo NT Ankle LDC Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zimmer Orthobiologics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSU2010-21B
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Defect of Articular Cartilage; Osteochondral Lesion of Talus; Osteochondritis Dissecans
Keywords: Talar injury; ankle; lesion; defect; cartilage repair
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DeNovo NT Subject: Subjects who have received or who are scheduled to receive a DeNovo NT Graft for repair of a cartilage lesion in the ankle.
  Interventions: Other: DeNovo NT Natural Tissue Graft

INTERVENTIONS:
Other: DeNovo NT Natural Tissue Graft — DeNovo NT is a juvenile cartilagenous tissue graft, inclusive of a viable human cartilage cells. It is provided as particulated tissue pieces of approximately 1mm3 each
  Other Names: DeNovo NT

SUMMARY:
The purpose of this post-market clinical study is to collect long-term outcomes for DeNovo NT Graft treatment of articular cartilage lesions in the ankle in a standard clinical setting. Outcomes to be assessed include pain, function, activity levels and healthcare resource use.

DETAILED DESCRIPTION:
Articular cartilage lesions in the ankle can cause significant pain and loss of function for young to middle age adults. There are several treatment options for symptomatic articular cartilage injuries depending on a patient's age, symptoms and duration of complaints in addition to the size and condition of the lesion. DeNovo NT Natural Tissue Graft is comprised of fresh particulated juvenile cartilage pieces that are secured inside articular cartilage lesions using fibrin adhesive. DeNovo NT Graft was developed due to the current need for expanded treatment options for the treatment of cartilage lesions, especially large lesions.

This post-market, multicenter, longitudinal data collection study was established to collect clinical outcomes of subjects implanted with DeNovo NT Graft. Data may be obtained either retrospectively or prospectively from patients implanted or to be implanted with DeNovo NT Graft for the treatment of lesion in the ankle. Data to be collected include details of the operative procedure as well as subject pain, function, activity levels, and healthcare resource use through a five year post-operative follow-up period.

ELIGIBILITY:
Potential subjects are screened for study entry based on a preliminary review of the inclusion and exclusion criteria as it applies to their pre-operative status (unless otherwise noted).

Inclusion Criteria:

* Has an articular cartilage lesion(s) in the ankle for which arthroscopic or surgical intervention with DeNovo NT Graft is warranted or has had prior treatment with DeNovo NT Graft for an articular cartilage lesion(s) in the ankle
* Has voluntarily signed the IRB approved informed consent
* Is of stable health and is able to undergo surgery
* Is male or female over the age of 18 at the time of consent
* Is physically and mentally willing and able to comply with post-operative rehabilitation and routinely scheduled clinical visits.

Exclusion Criteria:

* Displays a high surgical risk as determined by the investigative surgeon
* Is pregnant or breast-feeding
* Has a clinically diagnosed autoimmune disease
* Has an active joint infection or history of chronic joint infection at the surgical site
* Has medical history that would likely make the subject unreliable for the study, or any combination of variables in the investigator's judgment that should exclude a potential subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received or who are scheduled to receive a DeNovo NT graft for repair of a cartilage lesion in the ankle.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2011-03; Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Mean scores from patient-reported clinical outcome surveys | 5 years

SECONDARY OUTCOMES:
Incidence of reoperations and revision surgeries | 5 years

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, Davis at UC Davis Medical Center, Sacramento, California
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MedStar Health Research Institute at Union Memorial Hospital, Baltimore, Maryland
  - Minnesota Orthopedic Sports Medicine Institue at Twin Cities Orthopedics, Edina, Minnesota
  - OhioHealth Research Institute at Orthopedic Foot & Ankle Center, Westerville, Ohio
  - San Antonio Military Medical Center/Brooke Army Medical Center, Fort Sam Houston, Texas
  - The Orthopaedic Foot & Ankle Center of Washington, Falls Church, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Coetzee JC, Giza E, Schon LC, Berlet GC, Neufeld S, Stone RM, Wilson EL. Treatment of osteochondral lesions of the talus with particulated juvenile cartilage. Foot Ankle Int. 2013 Sep;34(9):1205-11. doi: 10.1177/1071100713485739. Epub 2013 Apr 10. PMID 23576118